CLINICAL TRIAL: NCT06948981
Title: A Single-arm, Open-label, Phase I/II Clinical Study of GT719 Injection for Recurrent/Refractory CD19 Positive Adult B-cell Malignancies
Brief Title: GT719 Injection for the Treatment of Recurrent/Refractory CD19 Positive Adult B-cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-001-056
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hematological Malignancy (Leukemia- Lymphoma)
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: GT719 Injection

INTERVENTIONS:
Biological: GT719 Injection — GT719 Injection

SUMMARY:
This study is a prospective single-arm open-labled phase I/II clinical trial, including dose escalation and expansion phase, aims to evaluate the safety, efficacy, and cellular pharmacokinetics of GT719 Injection in relapsed/refractory CD19 positive adult B-cell non Hodgkin lymphoma (B-NHL) and B-acute lymphoblastic leukemia (B-ALL) patients. A total of 46 subjects (anticipated) will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily enrolled in the study, signed an informed consent form, and willing and able to comply with the study protocol.

   -
2. Eastern Collaborative Oncology Group (ECOG) physical fitness status score of 0 or 1.

   -
3. CD19 positivity confirmed by flow cytometry and/or histopathology.

Exclusion Criteria:

1. Primary immunodeficiency.

   -
2. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to enrollment, requiring systemic anticoagulant therapy.

   -
3. Any medical condition that may interfere with the evaluation of the safety or effectiveness of research and treatment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events per CTCAE 5.0 | From infusion to the end of the treatment at 12 months
  To characterize the safety profile of GT719 in patients with recurrent/refractory CD19 positive adult B-cell malignant hematological tumor as measured by the incidence and severity of adverse events per CTCAE 5.0

SECONDARY OUTCOMES:
Objective response rate | 28 days post the first infusion, and follow-ups at Month 2, Month 3, Month 6, Month 9 and Month 12
  To evaluate efficacy parameters such as objective response rate(ORR) assessed by the Investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No